CLINICAL TRIAL: NCT06774352
Title: Prosthetic Breast Reconstruction After Mastectomy: Comparison of Clinical, Anthropometric and Patient Satisfaction Parameters
Brief Title: Prosthetic Breast Reconstruction After Mastectomy
Acronym: BrREC2020
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BrREC2020
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prosthetic breast reconstruction (DTI or EXP-IMPL): immediate prosthetic breast reconstructions (DTI - Direct to Implant) and in two surgical stages (EXP-IMPL - expander/prosthesis), after mastectomy

SUMMARY:
Breast cancer represents a disabling diagnosis for women, and the related destructive surgical intervention of mastectomy inevitably affects their social, relational and working life. The primary aim of post-oncological breast reconstruction is to restore volume, shape and projection as similar as possible to the contralateral breast, in unilateral mastectomies and between the two reconstructed breasts, in bilateral mastectomies, avoiding the patient the need to resort to uncomfortable and unsightly external prostheses.

The study in question has a purely observational and non-interventional nature, in order to evaluate whether today the traditional EXP-IMPL prosthetic reconstructive technique represents an obsolete option or whether it can still be considered a valid alternative in clinical, anthropometric and patient satisfaction terms

DETAILED DESCRIPTION:
The primary aim of post-oncological breast reconstruction is to restore volume, shape and projection as similar as possible to the contralateral breast, in unilateral mastectomies and between the two reconstructed breasts, in bilateral mastectomies, avoiding the patient the need to resort to uncomfortable and unexpectedly external prostheses.

The study in question has a purely observational and non-interventional nature, in order to evaluate whether today the traditional EXP-IMPL prosthetic reconstructive technique represents an obsolete option or whether it can still be considered a valid alternative in clinical, anthropometric and patient satisfaction terms. In order to evaluate outcomes in prosthetic breast reconstructions immediate (DTI - Direct to Implant) and in two surgical stages (EXP-IMPL - expander/prosthesis), after mastectomy, the aforementioned data will be subjected to appropriate statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Sex F
* Patients undergoing mastectomy (R-m, SS-m, NSS-m)
* Age 18 - 70
* Prosthetic breast reconstruction (DTI or EXP-IMPL)
* Written informed consent

Exclusion Criteria:

* Autologous breast reconstruction

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who underwent post-oncological prosthetic breast reconstruction in the period between 1.1.2011 - 31.5.2020, at the Plastic Surgery Unit of the University Hospital Company - Sant'Orsola Polyclinic - Bologna. The data recorded in the study derive from pre-operative and post-operative assessments, in accordance with daily clinical practice and normally performed for correct patient management.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | From the first patient entrolled, up to the 200th patient, an average of 2 years
  Technical Success is defined by number of reinterveions, major complication and the necessity to change approach.

SECONDARY OUTCOMES:
Patient satisfaction | From the first patient enrolled, up to the 200th. An average of 2 years
  Satisfaction is measured by specific Q-Breast questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Pinto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No